CLINICAL TRIAL: NCT02419092
Title: Investigation of Inflammation Induced by Obstructive Sleep Apnea: Effects of Continuous Positive Airway Pressure (CPAP), Massive Weight Loss and the Bioactive Compound Resveratrol
Brief Title: Obstructive Sleep Apnea-induced Changes in Adipose and Liver Tissue and Effects of Massive Weight Loss on Inflammation
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: LIRMOI-5-OSA
Record Dates: First submitted 2015-03-30; First posted 2015-04-17 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2016-01

CONDITIONS: Obesity; Obstructive Sleep Apnea
Keywords: Inflammation; Insulin resistance; Bariatric surgery
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive; Inflammation; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, urine, subcutaneous adipose tissue, visceral adipose tissue and liver tissue.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obstructive Sleep Apnea: Subjects scheduled to undergo bariatric surgery and with Obstructive Sleep Apnea
- No Obstructive Sleep Apnea, controls: Subjects scheduled to undergo bariatric surgery and without Obstructive Sleep Apnea, control group

SUMMARY:
UPDATED May 2016:

Originally the study design included investigation of the effects of the bioactive compound resveratrol compared to placebo tablets and to CPAP treatment. Due to fewer subjects having OSA than estimated by pre-study and, therefore, difficulties in the recruiting process the investigators have found it necessary to descale the study design. Hence, we have discontinued the resveratrol and CPAP intervention and will focus on the cross-sectional investigation of metabolic changes in subjects with and without OSA and the effect of weight loss after bariatric surgery on inflammation, OSA severity, metabolism and arterial stiffness.

Obstructive sleep apnea (OSA) is a common disorder especially among obese individuals and patients with type 2 diabetes. OSA is associated with an increased morbidity and mortality.

Continuous positive airway pressure (CPAP) is the standard treatment. Also weight loss is known to reduce the severity of OSA, especially bariatric surgery has proven effective because of the massive weight loss.

The investigators hypothesize that OSA via pro-inflammatory responses in various tissues causes low-grade inflammation which ultimately induce the associated co-morbidities. The investigators hypothesize that massive weight loss after bariatric surgery have beneficial effects on severity of OSA, inflammatory status and improves insulin sensitivity.

DETAILED DESCRIPTION:
UPDATED May 2016:

Originally the study design included investigation of the effects of the bioactive compound resveratrol compared to placebo tablets and to CPAP treatment. Due to fewer subjects having OSA than estimated by pre-study and, therefore, difficulties in the recruiting process the investigators have found it necessary to descale the study design. Hence, we have discontinued the resveratrol and CPAP intervention and will focus on the cross-sectional investigation of metabolic changes in subjects with and without OSA and the effect of weight loss after bariatric surgery on inflammation, OSA severity, metabolism and arterial stiffness.

OSA causes insulin resistance and seems to aggravate obesity related comorbidities such as hypertension, dyslipidemia and increase the risk of development of type 2 diabetes and non-alcoholic fatty liver disease.

More mechanisms may be involved in the pathogenesis of these negative effects from OSA but hypoxia-induced low-grade inflammation may play a central role since the levels of inflammatory markers generally are elevated in OSA. The tissues which are responsible for these systemic alterations are not known, however, adipose tissue might be a good candidate since it is known from studies that human adipose tissue can influence systemic inflammation.

Some studies even describe a small but significant anti-inflammatory effect and a beneficial effect on glucose metabolism following CPAP treatment. In addition, weight loss in patients with OSA is known to reduce the severity of or completely eliminate OSA.

The purpose of this study is primarily to investigate:

1. the metabolic changes in adipose and liver tissue induced by OSA in order to better understand how OSA negatively affects whole-body metabolism
2. the effect of weight loss after bariatric surgery on systemic inflammation, metabolism and the severity of OSA

24 subjects scheduled to undergo bariatric surgery will be recruited. They will all be screened for OSA. 12 subjects without OSA and 12 subjects with OSA will be included and examined before surgery and 6 months post-surgery.

The investigators will look at changes in:

* Inflammation-markers
* Biochemical markers of fat and sugar-metabolism
* Gene-expression in adipose and liver-tissue
* Severity of OSA
* Pulse-wave velocity

ELIGIBILITY:
Inclusion Criteria:

* Female/Male
* Legally competent (habil)
* 25-65 years old
* BMI > 35 and fulfill criteria for bariatric surgery in Denmark
* Written informed consent

Exclusion Criteria:

* Current treatment with CPAP
* Permanent treatment with glucocorticoids, NSAID or sleeping pills (otherwise discontinued for 1 week prior to inclusion)
* Severe heart, liver, kidney or lung disease
* Type 1 diabetes
* Work in transportation-related industry
* Pregnancy
* Substance abuse problem

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study groups will be selected from subjects referred to the outpatient clinics in Central Denmark Region and who meet the national guideline criteria for bariatric surgery.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Metabolic changes in adipose and liver tissue induced by OSA. Obese subjects with OSA will be compared to obese subjects without OSA. | Biopsies and blood samples obtained in relation to bariatric surgery
  Cross-sectional genetic and metabolic analysis of biopsies and blood samples obtained in relation to bariatric surgery on subjects with and without sleep apnea. In tissue samples gene-expression profile is measured using Affymetrix gene array and blood samples are used for metabolic profiling and inflammatory markers (hs-CRP, TNFalfa, IL-6, IL-8, adiponectin, leptin, MCP-1, FGF211, CD163)

SECONDARY OUTCOMES:
Effect of bariatric surgery on adipose tissue inflammation and systemic inflammation. | Evaluated at time of bariatric surgery and at follow-up 6 months after bariatric surgery.
  Changes in inflammation markers (hs-CRP, TNFalfa, IL-6, IL-8, adiponectin, leptin, MCP-1, FGF21, CD163) in blood and adipose tissue.
  Changes in expression of mRNA of the relevant inflammatory pathways assessed by gene expression studies.
Effect of bariatric surgery on insulin sensitivity. | Evaluated at time of bariatric surgery and at follow-up 6 months after bariatric surgery
  Changes in insulin sensitivity assessed by HOMA-IR, fructosamine and correction in oral anti diabetic medication.
Effect of bariatric surgery on the severity of OSA. | Evaluated at baseline, 4 weeks post-bariatric surgery and 6 months post-bariatric surgery
  Changes in AHI-score and Sleepiness Score (based on questionnaires).

OTHER OUTCOMES:
Arterial stiffness assessed by office carotid-femoral pulse-wave | Evaluated at baseline, end of intervention and 6 months post-bariatric surgery
  Changes in arterial stiffness assessed by office carotid-femoral pulse-wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Steen B Pedersen, MD,Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: Undecided